CLINICAL TRIAL: NCT04762992
Title: Low Molecular Weight Heparin for the Treatment of Early Fetal Growth Restriction
Brief Title: LMWH for Treatment of Early Fetal Growth Restriction (HepaGrowth)
Acronym: HepaGrowth
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Centro Hospitalar de Lisboa Central (Other)
Collaborators: NOVA Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHULC.CI.452.2018
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-03

CONDITIONS: Fetal Growth Retardation; Prematurity; Pre-Eclampsia
Keywords: Fetal Growth Retardation; Prematurity; Pre-Eclampsia; Placenta
MeSH Terms: conditions — Fetal Growth Retardation; Premature Birth; Pre-Eclampsia | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: pharmacological intervention and standard of care arms
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Blinded to clinicians performing the ultrasound and outcomes assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group, enoxaparin (Experimental): Enoxaparin subcutaneous injections
  Interventions: Drug: subcutaneous Enoxaparin
- Standard of care (Other): Obsteric standard of care
  Interventions: Other: standard of care

INTERVENTIONS:
Drug: subcutaneous Enoxaparin — Enoxaparin subcutaneous injections (40 mg, 4000 IU daily) starting immediately after the diagnosis of FGR, and until 36 weeks of gestation or 12 hours before delivery, whichever comes first.
  Other Names: experimental
  Arms: Intervention group, enoxaparin
Other: standard of care — Obsteric standard of care.
  Arms: Standard of care

SUMMARY:
Early fetal growth restriction (FGR) is associated with considerable fetal and neonatal morbimortality. Placental thrombosis, infarcts and hypercoagulability are frequently seen in these pregnancies, suggesting a role for the activation of the coagulation cascade in the genesis of FGR. Patients will be randomized for low-molecular weight heparin or standard of care, and the outcomes of both arms (gestational age at delivery, gestational and fetal morbidity) will be compared.

DETAILED DESCRIPTION:
FGR is the second leading cause of perinatal mortality, being associated with approximately 30% of stillbirths. Early FGR is associated with substantial disturbances of placental implantation and fetal hypoxia, which requires fetal cardiovascular adaptation. Both maternal and fetal Doppler alterations are present, allowing for risk stratification and monitoring. Although the precise etiology for FGR due to placental causes is unknown, placental thrombosis, infarcts and hypercoagulability are frequently seen, suggesting a role for the activation of the coagulation cascade in the genesis of FGR. Currently, the management of early FGR is limited to the monitoring of fetal Doppler parameters until the risks for preterm delivery outweight the benefits of ongoing monitoring. As such, there is a special need for effective preventive and therapeutic interventions that improve the outcomes. Low molecular weight heparin (LMWH), for its anticoagulant and anti-inflammatory properties has been suggested as a possible therapeutic agent in this setting. The investigators will randomize the participants to two intervention arms in a one-to-one ratio, using a computer generated randomization program. The randomization will be stratified for gestational age at diagnosis of FGR (22 to 26 weeks and >26 to 32 weeks). The experimental group will be administered enoxaparin subcutaneous injections (40 mg, 4000 IU daily) and the control group will be provided standard of care. Both groups will start intervention immediately after the diagnosis of FGR, and will continue it until 36 weeks of gestation or 12 hours before delivery, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. being 18 years old or older
2. being able to provide consent
3. having a viable singleton pregnancy with diagnosed early FGR confirmed in our unit according to the 2020 International Society of Ultrasound in Obstetrics & Gynecology (ISUOG) criteria (one solitary parameter: estimated fetal weight/ abdominal circumference lower than the 3rd centile or absent end-diastolic flow in umbilical artery; or estimated fetal weight/abdominal circumference below the 10th centile combined with either umbilical artery pulsatility index > 95th centile or uterine artery mean pulsatility index > 95th centile)

Exclusion Criteria:

1. multiple gestation;
2. diagnosed fetal chromosomal abnormalities;
3. associated fetal morphological malformations;
4. evidence of fetal infection (serological or after invasive testing);
5. use of LMWH or NFH in the index pregnancy before randomization or start of any of these medications for another indication if the patient is in the control group
6. present use of systemic salicylates in anti-inflammatory dosage (> 150mg/day) or NSAIDs (including ketorolac)
7. maternal history of allergy to LMWH or non-fractionated heparin (NFH);
8. hypersensitivity to pork products;
9. maternal history of heparin-induced thrombocytopenia;
10. maternal thrombocytopenia (platelets < 100 000);
11. history of maternal hemophilia or Von Willebrand disease
12. presence of placental hematoma;
13. maternal diabetic retinopathy;
14. bacterial endocarditis;
15. active clinically significant bleeding and conditions with a high risk of hemorrhage, including recent hemorrhagic stroke, gastrointestinal ulcer, presence of malignant neoplasm at high risk of bleeding, recent brain, spinal or ophthalmic surgery, known or suspected esophageal varices, arteriovenous malformations, vascular aneurysms or major intraspinal or intracerebral vascular abnormalities;
16. persistent blood pressure > 160/100 mmHg, despite optimal anti-hypertensive regimen;
17. history of severe renal disease (eGFR <30mL/min);
18. known or suspected hepatic impairment;
19. current participation in another clinical trial;
20. patients that are not part of the national health system (SNS);
21. delivery already scheduled, or predicted in the next 7 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — biologic (genotipic and fenotipic) female sex
Enrollment: 12 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Gestational age at delivery | day of delivery
  Best assessment of the time of gestation, either by first trimester sonography, last menstrual day or day of implantation of in vitro conception product

SECONDARY OUTCOMES:
Neonatal birtweight and birthweight centile | day of delivery
  Weight at birth of the newborn (in grams) and respective percentile
Newborn Apgar Score in the 5th minute | day of delivery
  Newborn Apgar score in the 5th minute, assessed by a nurse or pediatrician
Newborn Umbilical Artery pH | day of delivery
  pH of the umbilical artery, assessed immediately after delivery
Stillbirth, neonatal intensive care admission and duration of admission | from randomization up to 1 year after delivery
  A composite outcome of severe neonatal morbidity (evidence of one or more of: intraventricular hemorrhage grade 3 or 4; cystic periventricular leukomalacia; chronic lung disease; retinopathy of prematurity requiring treatment; necrotizingenterocolitis requiring surgery
Maternal and fetal Doppler parameters | from randomization to delivery
  Pulsatility index (PI) of the uterine arteries, PI anddiastolic flow in the umbilical artery, PI in the middle cerebral artery, cerebro-placental ratio, ductusvenosus PI and a wave
Placental pathology | day of delivery
  Percentage of placenta occupied by fibrosis or infarcts
Sflt1-PLGF ratio | from randomization to delivery
  Evolution of Sflt1-PLGF ratio from diagnosis of FGR to delivery
Syncytiotrophoblast membrane extracellular vesicles (STB-EV) | from randomization up to 1 week after delivery
  Protein and genetic composition
Gestational hypertension or preeclampsia; placental abruption | from randomization up to 1 week after delivery
  Pregnancy induced hypertension, preeclamspia,HELLP syndrome
Antepartum hemorrhage; maternal thrombocytopenia (platelets < 100 000 x 10 9/L); postpartum hemorrhage | from randomization up to 1 week after delivery
  Hemorrhage, bruising,pain
Mode and indication for delivery | from randomization up to 48h after delivery
  As spontaneous vaginal birth, operative vaginal birth (forceps orvacuum/ventouse), or cesarean section. For induced labor or planned cesarean section, theindication for scheduling the delivery will be documented (e.g., gestational age, maternal or fetalindications). In cases of operative vaginal or cesarean delivery, the indication for intervention willbe specified (e.g., non-reassuring fetal status, labor dystocia).

CONTACTS AND LOCATIONS:
Overall Officials: Fátima Serrano, MD, PhD, Study Chair — Centro Hospitalar Universitário de Lisboa Central; Catarina Palma-dos-Reis, MD, MSc, Principal Investigator — Centro Hospitalar Universitário de Lisboa Central
Locations (1):
- Centro de Diagnóstico Pré-Natal, Maternidade Dr. Alfredo da Costa, Centro Hospitalar Universitário de Lisboa Central, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller J, Turan S, Baschat AA. Fetal growth restriction. Semin Perinatol. 2008 Aug;32(4):274-80. doi: 10.1053/j.semperi.2008.04.010. PMID 18652928
- [Background] Nardozza LMM, Zamarian ACP, Araujo Junior E. New Definition of Fetal Growth Restriction: Consensus Regarding a Major Obstetric Complication. Rev Bras Ginecol Obstet. 2017 Jul;39(7):315-316. doi: 10.1055/s-0037-1603741. Epub 2017 Jun 12. No abstract available. PMID 28605820
- [Background] Arbeille P, Maulik D, Fignon A, Stale H, Berson M, Bodard S, Locatelli A. Assessment of the fetal PO2 changes by cerebral and umbilical Doppler on lamb fetuses during acute hypoxia. Ultrasound Med Biol. 1995;21(7):861-70. doi: 10.1016/0301-5629(95)00025-m. PMID 7491742
- [Background] Nardozza LM, Caetano AC, Zamarian AC, Mazzola JB, Silva CP, Marcal VM, Lobo TF, Peixoto AB, Araujo Junior E. Fetal growth restriction: current knowledge. Arch Gynecol Obstet. 2017 May;295(5):1061-1077. doi: 10.1007/s00404-017-4341-9. Epub 2017 Mar 11. PMID 28285426
- [Background] Elder MG, Myatt L. Coagulation and fibrinolysis in pregnancies complicated by fetal growth retardation. Br J Obstet Gynaecol. 1976 May;83(5):355-60. doi: 10.1111/j.1471-0528.1976.tb00842.x. PMID 1268144
- [Background] Bellart J, Gilabert R, Fontcuberta J, Carreras E, Miralles RM, Cabero L. Coagulation and fibrinolytic parameters in normal pregnancy and in pregnancy complicated by intrauterine growth retardation. Am J Perinatol. 1998 Feb;15(2):81-5. doi: 10.1055/s-2007-993903. PMID 9514130
- [Background] Fuke Y, Aono T, Imai S, Suehara N, Fujita T, Nakayama M. Clinical significance and treatment of massive intervillous fibrin deposition associated with recurrent fetal growth retardation. Gynecol Obstet Invest. 1994;38(1):5-9. doi: 10.1159/000292434. PMID 7959327
- [Background] Seravalli V, Baschat AA. A uniform management approach to optimize outcome in fetal growth restriction. Obstet Gynecol Clin North Am. 2015 Jun;42(2):275-88. doi: 10.1016/j.ogc.2015.01.005. PMID 26002166
- [Background] Tyrell DJ, Kilfeather S, Page CP. Therapeutic uses of heparin beyond its traditional role as an anticoagulant. Trends Pharmacol Sci. 1995 Jun;16(6):198-204. doi: 10.1016/s0165-6147(00)89022-7. PMID 7652929
- [Background] Lewander R, Lunell NO, Nylund L, Sarby B, Thornstrom S. [Uterine-placental blood flow. Method of measurement and clinical use]. Lakartidningen. 1980 Jan 30;77(5):333-4. No abstract available. Swedish. PMID 7366291
- [Background] Seravalli V, Block-Abraham DM, Turan OM, Doyle LE, Blitzer MG, Baschat AA. Second-trimester prediction of delivery of a small-for-gestational-age neonate: integrating sequential Doppler information, fetal biometry, and maternal characteristics. Prenat Diagn. 2014 Nov;34(11):1037-43. doi: 10.1002/pd.4418. Epub 2014 Jun 11. PMID 24864018
- [Background] Picklesimer AH, Oepkes D, Moise KJ Jr, Kush ML, Weiner CP, Harman CR, Baschat AA. Determinants of the middle cerebral artery peak systolic velocity in the human fetus. Am J Obstet Gynecol. 2007 Nov;197(5):526.e1-4. doi: 10.1016/j.ajog.2007.04.002. PMID 17980196
- [Result] Yu YH, Shen LY, Zou H, Wang ZJ, Gong SP. Heparin for patients with growth restricted fetus: a prospective randomized controlled trial. J Matern Fetal Neonatal Med. 2010 Sep;23(9):980-7. doi: 10.3109/14767050903443459. PMID 19951008
- [Result] Yu YH, Shen LY, Zhong M, Zhang Y, Su GD, Gao YF, Quan S, Zeng L. [Effect of heparin on fetal growth restriction]. Zhonghua Fu Chan Ke Za Zhi. 2004 Dec;39(12):793-6. Chinese. PMID 15733401